CLINICAL TRIAL: NCT07072520
Title: A Pilot Study on the Association of Dietary Inflammatory Index and Healthy Eating Index-2015 With Body Composition in Female Nutrition and Dietetics Students
Brief Title: Diet Quality and Body Composition in Female Students
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Rahime Evra KARAKAYA, Principal Investigator, Ankara Yildirim Beyazıt University
Other Study IDs: AnkaraYBU-KARAKAYA006
Record Dates: First submitted 2025-07-07; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Female
Keywords: diet quality; inflammation; body composition; female
MeSH Terms: conditions — Inflammation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- University students: Female university students
  Interventions: Behavioral: Questionnaire; Other: Body composition assessment

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire including sociodemographic characteristics and dietary assessment
Other: Body composition assessment — Body Composition Assessment via bioelectrical impedance analysis (BIA)

SUMMARY:
The goal of this observational study is to learn about the relationship between diet quality and body composition in female university students. The main question it aims to answer is:

Is there a relationship between diet quality and body composition in female university students?

Participants will answer survey questions about sociodemographic characteristics. 24 hour dietary recalls will be taken to evaluate diet quality. Body composition will be assessed via Bioelectrical impedance analysis (BIA).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Nutrition and Dietetics student
* Age: 19-30 years

Exclusion Criteria:

* Pregnant or lactating
* Individuals with a pacemaker

Ages: 19 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University students
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Dietary Inflammatory Index | Baseline
  The Dietary Inflammatory Index (DII) is a literature-derived scoring system that assesses the inflammatory potential of an individual's diet based on the intake of various nutrients and food components. Higher scores indicate a more pro-inflammatory diet, while lower scores indicate an anti-inflammatory one.
Healthy eating index-2015 | Baseline
  The Healthy Eating Index-2015 (HEI-2015) is a measure developed by the U.S. Department of Agriculture to assess how well an individual's dietary intake aligns with the 2015-2020 Dietary Guidelines for Americans. Scores range from 0 to 100, with higher scores indicating better adherence to dietary recommendations. Specifically, a score above 80 reflects "good" diet quality, scores between 51 and 80 suggest "moderate" quality, while scores of 50 or below are classified as "poor" diet quality.

SECONDARY OUTCOMES:
Body fat | Baseline
  Body fat mass in kg
Body fat | Baseline
  Body fat in percentage (%)
Fat free mass | Baseline
  Fat free mass in kg
Skeletal muscle mass | Baseline
  Skeletal muscle mass in kg
Total body water | Baseline
  Total body water in kg
Total body water | Baseline
  Total body water in percentage (%)
Phase angle | Baseline
  Phase angle in degrees
Body weight | Baseline
  Body weight in kg
Height | Baseline
  Height in cm

CONTACTS AND LOCATIONS:
Overall Officials: Rahime E Karakaya, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Çubuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No